CLINICAL TRIAL: NCT06055699
Title: Association Between the Occurrence of a Clinical RElapse and Gut MIcrobiota Modifications: a Cohort Study of Patients With pSOriasis
Acronym: REMISSIOn
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP230758
Record Dates: First submitted 2023-09-20; First posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Psoriasis; Microbial Colonization
Keywords: microbiota; pSOriasis; anti-IL17 biologic agents; anti-IL23 biologic agents
MeSH Terms: conditions — Psoriasis; Communicable Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool samples are a collection of products derived from the human body that is not invasive in any way and samples not taken as part of usual care. Stool samples will be collected at home within 7 days of the visit M0, M3 and M6 and within 14 days of the visit M12
  Blood samples (serum, 15 ml) are an additional and minimal collection performed following a sample taken as part of usual care. Blood samples (serum) will be collected during the visit at M0, M3 (± 7 days), M6 (± 7 days) and M12 (± 7 days).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with psoriasis in remission: Patients with psoriasis in remission after IL23i or IL17inhibitor treatments and who have stopped their medication for 2 to 4 weeks.
  Interventions: Other: Fecal sampling; Other: Blood sampling

INTERVENTIONS:
Other: Fecal sampling — Stool samples are a collection of products derived from the human body that is not invasive in any way and samples not taken as part of usual care.
  Stool samples will be collected at home within 7 days of the visit M0, M3 and M6 and within 14 days of the visit M12 in an ethanol tube and in DNA/RNA shield, and transported at room temperature to Saint-Antoine Hospital (CRB SAT, AP-HP, Pr. SIMON ), samples will be aliquoted (3 aliquots per tubes) and stored at -80°C for a period of 5 years (renewable) At the end of the research, stool samples will be analysed using metagenomics sequencing.
  DNA extraction will be performed following the standards of the The International Human Microbiome Standards . DNA will be stored at -80°C.
  Other Names: Stool samples
Other: Blood sampling — Blood samples (serum, 15 ml) are an additional and minimal collection performed following a sample taken as part of usual care.
  Blood samples (serum) will be collected during the visit at M0, M3 (± 7 days), M6 (± 7 days) and M12 (± 7 days).
  In the hours following collection, the samples must be aliquoted and stored at -80°C in a secure place in the participating centre.
  Other Names: Blood samples (serum)

SUMMARY:
The human microbiota corresponds to an extremely rich and varied set of microorganisms that colonize our various epitheliums from birth, including the intestine, lungs and skin, where they interact continuously with our immune system. Changes in microbial composition and function, termed dysbiosis, have been linked to alterations in immune responses and to disease development, such as psoriasis. Recent research has shown that the gut microbiota can condition the therapeutic response to checkpoint inhibitors and that fecal microbiota transplant overcomes resistance to these therapy, suggesting a direct role for the microbiota in the ability to shape a therapeutic immune response. Antibiotic exposure during the course of cancer therapy negatively correlates with patients' response to anti-PD-1 treatment response, thus highlighting the link between the enrichment of specific microbial taxa in intestines and the response to immunotherapy. This observation suggests that treatments capable of modulating microbial networks and promoting specific bacterial clades may modulate the host's immune response. Hence, beyond their expected effect in the targeted tissue, part of the therapeutic effect of drugs could rely on this mechanism. In psoriasis patients, observational studies suggest that gut microbiome is altered differently after the use of anti-IL17 or anti-IL23 biologic agents.

Main objective: To determine the evolution of microbial composition of fecal samples issued to patients who responded to a biologic agent (IL-17 inhibitors, IL-23 inhibitors) and have stopped their treatment for 2 to 4 weeks before the index date, at baseline and 6 months or clinical relapse after treatment discontinuation

Design of the study: Prospective french multicentre observational cohort study

Population of study participants: Patients with psoriasis in remission after IL23i or IL17inhibitor treatments and who have stopped their medication for 2 to 4 weeks.

Number of participants included: 50 adult patients considered in remission and have stopped for at least 2 weeks and a maximum of 4 weeks, one of the following biologic agent: secukinumab, ixekizumab, brodalumab, bimekizumab, guselkumab, tildrakizumab, or risankizumab

ELIGIBILITY:
Inclusion Criteria:

* Subject over 18 years of age
* Subject diagnosed with psoriasis considered in remission (as defined by absolute PASI<2 within 6 months of follow-up)
* Subject who has stopped his biologic agent including IL-17 inhibitors or IL-23 inhibitors for 2 to 4 weeks.
* Written informed consent for participation in the study

Exclusion Criteria:

* Subject currently experiencing or having a history of other concomitant skin conditions that would interfere with evaluation of psoriasis
* Subject treated by NSAIDs, antibiotics, antifungals, antivirals or proton-pump inhibitors within 4 weeks before inclusion (or foreseeable use during the study)
* Subject with a concomitant diagnosis of cirrhosis, coeliac disease or signs of bacterial infection
* Subject has concurrent acute or chronic viral hepatitis B or C or human immunodeficiency virus (HIV) infection
* Subject having a personal or familial history of psoriatic arthritis or inflammatory bowel disease
* Subject with BMI<18.5 or BMI>35
* Subject consuming probiotics or using specific diet with many dietary exclusions according to the discretion of the investigator
* Pregnant and /or breastfeeding woman,
* Subject deprived of liberty by judicial or administrative decision or patient under guardianship
* Subject unable to understand the purpose and conditions of the study and unable to give consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with psoriasis in remission after IL23i or IL17inhibitor treatments and who have stopped their medication for 2 to 4 weeks.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Microbial features | after 6 months of the baseline visit or the first occurrence of psoriasis clinical relapse after baseline visit
  Microbial features (gene richness, species, functional modules) impacted by the discontinuation of the biologic agent after 6 months or the first occurrence of psoriasis clinical relapse.

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Sbidian, MD-PhD, Principal Investigator — APHP

IPD SHARING:
Plan to Share IPD: No